CLINICAL TRIAL: NCT01962077
Title: Comparison of MedCem MTA and Formocresol Used in Pulpotomies in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nathalie- HMO-CTIL
Record Dates: First submitted 2013-09-25; First posted 2013-10-14 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Pulpotomies Primary Teeth; Effectiveness of MedCem MTA® in Pulpotomies Primary Teeth
Keywords: pulpotomy; MTA; primary teeth; formocresol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MedCem MTA pulpotomies (Experimental)
  Interventions: Procedure: MedCem MTA pulpotomies in primary teeth.

INTERVENTIONS:
Procedure: MedCem MTA pulpotomies in primary teeth.

SUMMARY:
assess the effect of MedCem MTA as a pulp medicament following pulpotomy in human primary molars with carious pulp exposure in comparison to Formocresol.

ELIGIBILITY:
Inclusion Criteria:

1. healthy children
2. with Asymptomatic primary molars with a deep carious lesion;
3. Exposure of a vital pulp by caries;
4. No clinical or radiographic evidence of pulp degeneration, such as excessive bleeding from the root canal, internal root resorption, inter-radicular and/or periapical bone destruction,swelling, or sinus tract;
5. Ability to perform a leakage free restoration of the teeth using stainless steel crown, or amalgam/resin based restoration.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Success of MedCem MTA pulpotomy in primary molar | Up to 36 months
  No pain, no swelling or sinus tract, no internal root resorption progressing into the bone, no furcation and/or periapical bond destruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel